CLINICAL TRIAL: NCT05868460
Title: Impact of High Intensity Laser Therapy on Temporomandibular Joint Disorders After Head and Neck Cancer.
Brief Title: Laser Therapy on TMJ Disorders After Head and Neck Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004499
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2023-05

CONDITIONS: Temporomandibular Joint Disorders
Keywords: High Intensity Laser Therapy; Temporomandibular Joint Disorders; Head And Neck Cancer
MeSH Terms: conditions — Temporomandibular Joint Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (High Intensity Laser Therapy Group) (Experimental): patients will receive HILT in addition to traditional physical therapy exercise program
  Interventions: Device: High intensity laser; Other: traditional physical therapy exercise program
- Group B (Placebo-Control Group) (Placebo Comparator): patients will receive placebo HILT in addition to traditional physical therapy exercise program
  Interventions: Other: traditional physical therapy exercise program; Device: placebo High intensity laser

INTERVENTIONS:
Device: High intensity laser — patients will receive Nd: YAG with wavelength 1064 nm, peak power 3KW, energy density 360-1780 mJ/cm2, a short duration 120-150 micro sec, a mean power 10.5 W, a low frequency 10-40 HZ, a duty cycle of 0.1%, a probe diameter of 0.5 cm and spot size of 0.2 cm2. The treatment will be applied into 3 phases in each session. In addition to the traditional physical therapy exercise program (passive and active ROM exercises, stretching and strengthening exercises) for 20 minutes, total session time is 35 minutes, 3 days/ week for 4 weeks.
  Arms: Group A (High Intensity Laser Therapy Group)
Other: traditional physical therapy exercise program — passive and active ROM exercises, stretching and strengthening exercises for 35 minutes, 3 days/ week for 4 weeks.
Device: placebo High intensity laser — patients will receive placebo HILT including the same treatment as in group A but the laser device will be turned off.
  Arms: Group B (Placebo-Control Group)

SUMMARY:
Temporomandibular disorder (TMD) is a term describing musculoskeletal conditions of the face, jaw and temporal regions. TMD is frequently associated with pain and/or dysfunction such as impaired jaw function, pain in the temporomandibular joint (TMJ), muscles and/or related structures, and associated headaches. The aetiology of TMD is multifactorial and complex.

DETAILED DESCRIPTION:
It is known that one cause of TMD symptom development is treatment for head and neck cancer (HNC). The main treatment modalities for HNC include radiotherapy (RT) with or without chemotherapy and surgical intervention, either as a single therapy or a combination therapy. In the head and neck region, the anatomical structures are necessary for essential functions such as speech, swallowing, breathing, smell, and taste. The treatment of head and neck tumours may frequently impair some of these functions, which may result in pain, oral dysfunction, and impaired health-related quality of life.

High intensity laser therapy (HILT) is a non-invasive and painless treatment method. The latest studies have reported the beneficial effects of neodymium-doped yttrium aluminum garnet (Nd: YAG) laser therapy in patients with pain. The advantage of HILT over low level laser therapy (LLLT) is that HILT is able to penetrate and stimulate wider and/or deeper areas; thus, considerably more energy may be transmitted to tissue during HILT therapy compared to LLLT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with temporomandibular joint disorders (myofascial pain, trismus and limitation of ROM) after head and neck cancer, patients will be diagnosed by an experienced oral and maxillofacial surgeon.
2. Patients with 20 to 60 years old.
3. 6 months after ending radiotherapy.

Exclusion Criteria:

1. Patients with implants.
2. Current metastasis.
3. Continuing radiotherapy.
4. Pregnant females.
5. Sensitivity to phototherapy.
6. Bells palsy.
7. Subjects with disk displacement, arthralgia or osteoarthritis at TMJ.
8. Subjects who received analgesics or antidepressants.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  It will be measured by visual analogue scale. It starts with no pain at the left side and gradually increasing pain towards the end of the line at the right side (0-10) and high scores indicate greater pain.

SECONDARY OUTCOMES:
Range of motion | 4 weeks
  Range of motion of temporomandibular joint will be measured by Vernier caliper scale
Muscle power assessment | 4 weeks
  Surface electromyography (EMG) will be used to evaluate the strength of the masseter and anterior temporal muscles
Functional disability | 4 weeks
  It will be measured by jaw functional limitation scale-20. It has a score range of 1 to 200, and high scores indicate worsening jaw function.
Quality of life (Oral health Impact Profile) | 4 weeks
  By using the Oral health Impact Profile consisted of 7 different domains (functional limitation, physical pain, psychological discomfort, psychological disability, physical disability, social disability, and handicap). Each domain was assessed by two questions, scored using a 5-point Likert scale (0 = never to 4 = very often). The total score was derived by a summing of the domain scores, it can range from 0 to 56. A higher score indicates a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hadaya M Eladl, PhD, Study Director — Assisstant professor of physical therapy for surgery, Faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: Study protocol